CLINICAL TRIAL: NCT00281437
Title: Health First: Health and Psychological Outcomes of Physical Activity- Study 2
Brief Title: Health First-Study 2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0503-03
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Exercise Adherence; Sedentary Adults; Lifestyle; Traditional
Keywords: exercise; adherence; lifestyle; choice; autonomy
MeSH Terms: conditions — Motor Activity

INTERVENTIONS:
Behavioral: choice of exercise program

SUMMARY:
The current study was designed to investigate the influence of choice of exercise program on exercise adherence. The two exercise programs included 1) traditional exercise at a fitness centre or 2) lifestyle exercise-walking using a pedometer to track steps. Biological and psychological indicators were examined to investigate the effect of choice in a sample of sedentary adults.

ELIGIBILITY:
Inclusion Criteria:

* 25-65 year old adults
* sedentary (exercise less than twice per month in the last 4 months)

Exclusion Criteria:

* physician non-consent
* too active (exercise more than twice per month in the last 4 months)
* participated in previous studies from this lab

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Rodgers, PhD, Principal Investigator — University of Alberta; Gordon J Bell, PhD, Principal Investigator — University of Alberta; Kerry Courneya, PhD, Principal Investigator — University of Alberta; Vicki J Harber, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada